CLINICAL TRIAL: NCT02017886
Title: Salivary IgA and Cytokines Response to Dietary Supplementation of Lactobacillus Reuteri
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Copenhagen (Other)
Responsible Party: Principal Investigator, Mette Rose Jørgensen, PhD-student, dentist, University of Copenhagen
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: H-4-2013-158
Record Dates: First submitted 2013-12-04; First posted 2013-12-23 (Estimated); Last update posted 2016-05-11 (Estimated); Status verified 2016-05

CONDITIONS: Dental Caries; Periodontitis
Keywords: Probiotics; Oral health; Innate immunity
MeSH Terms: conditions — Dental Caries; Periodontitis

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- L. reuteri DSM 17938/ATCC PTA (Active Comparator): L. reuteri DSM 17938/ATCC PTA twice daily for three weeks.
  Interventions: Dietary Supplement: L. reuteri DSM 17938/ATCC PTA
- Placebo (Placebo Comparator): Placebo tablet twice daily for three weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: L. reuteri DSM 17938/ATCC PTA — L. reuteri DSM 17938/ATCC PTA twice daily for three weeks
  Arms: L. reuteri DSM 17938/ATCC PTA
Dietary Supplement: Placebo — Placebo tablet twice daily for three weeks
  Arms: Placebo

SUMMARY:
To evaluate the effect of daily ingestion of the probiotic Lactobacillus reuteri on the levels of secretory IgA and the cytokines Il1-beta, IL-6, IL-8 and IL-10 in saliva of healthy young adults.

DETAILED DESCRIPTION:
Study design: A randomized, double-blind, cross-over design separated by three weeks run-in and wash-out periods. Each intervention period is three weeks and the participants are allocated to the test and placebo regimes in a randomized order.

Material: 41 healthy adults are enrolled after informed consent from the School of Dentistry, University of Copenhagen.

Methods: Samples of resting, unstimulated whole saliva (UWS) and stimulated whole saliva (SWS) are collected five times during the study period. The samples are immediately frozen in 0.5 ml aliquots.

Intervention: The subjects are instructed to ingest two tablets containing Lactobacillus reuteri or placebo, twice daily for 3 weeks. No probiotic food or health products are allowed during the intervention period. All normal oral hygiene routines should be maintained during the entire study. The compliance is checked through interviews. Any perceived side effects are reported without delay to the research staff.

Endpoints: The concentration of total protein and secretory IgA in saliva are determined with the enzyme-linked immune-sorbent assay (ELISA). The levels of the cytokines IL1-beta, IL-6, IL-8 and IL-10 is determined by Luminex-technology.

Scientific importance: The study may provide evidence that probiotic supplements can influence the innate defense system in the whole saliva which may open up for novel strategies to combat oral diseases.

ELIGIBILITY:
Inclusion Criteria:

* Healthy individuals with no chronic compromising illnesses
* No medication intake for serious chronic diseases
* No regular intake of probiotic products up till one month before inclusion

Exclusion Criteria:

* Recent antibiotic therapy (within the last six months)
* Pregnant or lactating women
* Active infection that needs treatment with antibiotics

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2013-11; Primary Completion 2015-12 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
The overall aim of this study is to evaluate the effect of daily ingestion of Lactobacillus reuteri on the levels of secretory IgA and cytokines in whole saliva of healthy adults. | Participants will be followed for 12 weeks after inclusion. Saliva samples will be analyzed and data presented when all 40 participants have completed the intervention period.
  Endpoints: The concentration of total protein and secretory IgA in saliva are determined in duplicates with the Bio-Rad protein assay and enzyme-linked immune-sorbent assay (ELISA), respectively. Values are express as mg/100ml or %IgA/protein.

CONTACTS AND LOCATIONS:
Overall Officials: Mette Rose Jørgensen, PhD-student, Principal Investigator — University of Copenhagen
Locations (1):
- University of Copenhagen, Copenhagen, Kbh. N, Denmark

REFERENCES:
- [Derived] Jorgensen MR, Keller MK, Kragelund C, Hamberg K, Ericson D, Nielsen CH, Twetman S. Lactobacillus reuteri supplements do not affect salivary IgA or cytokine levels in healthy subjects: A randomized, double-blind, placebo-controlled, cross-over trial. Acta Odontol Scand. 2016 Jul;74(5):399-404. doi: 10.3109/00016357.2016.1169439. Epub 2016 Apr 22. PMID 27104984